CLINICAL TRIAL: NCT00345540
Title: Phase 2 Trial of NOV-002 With Carboplatin in Women With Recurrent and Platinum Resistant Tumors of Mullerian Origin
Brief Title: Efficacy of NOV-002 in Combination With Carboplatin in Chemotherapy-resistant Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Collaborators: Massachusetts General Hospital (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV002- IS21 -OC
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2009-01

CONDITIONS: Ovarian Cancer
Keywords: Platinum Resistant Tumors of Ovarian Origin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — NOV 002; Glutathione Disulfide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOV-002 plus Carboplatin (Experimental): NOV-002 is given by IV bolus on lead-in day -1 at cycle 1, and on day 1 at subsequent cycles, followed by Carboplatin AUC 5. NOV-002 is then continued via daily SC injection, with 28 day cycles.
  Interventions: Drug: NOV-002; Drug: Carboplatin

INTERVENTIONS:
Drug: NOV-002 — 60 mg / mL / day / 20-23 Days
  Other Names: Oxidized Glutathione
Drug: Carboplatin — AUC 5 following IV bolus administration of NOV-002
  Other Names: Paraplatin

SUMMARY:
The purpose of this trial is to determine the tumor response rate of NOV-002 plus carboplatin in a cohort of women with platinum resistant cancer of ovarian origin.

DETAILED DESCRIPTION:
The purpose of this research study is to learn if adding NOV-002 to the chemotherapy drug carboplatin works in treating ovarian cancer. Platinum containing drugs such as carboplatin are the standard treatment for ovarian cancer, and are effective for many women. However, in many women the cancer eventually stops responding to the chemotherapy (becomes resistant).

The active part of NOV-002 is a substance made by the body that is involved in many chemical reactions in cells. NOV-002 does not directly kill cancer cells, but previous research has shown that it may make cancer cells more likely to be killed by chemotherapy drugs. Specifically, it may help platinum chemotherapy kill cancer that has become resistant to platinum chemotherapy. Previous trials have also shown that patients receiving NOV-002 in addition to carboplatin may have tolerated chemotherapy better than those who received chemotherapy alone. NOV-002 has been used in other research studies on various types of cancer. It is approved for use in Russia. It is not approved by the US Food and Drug Administration (FDA) for use outside of research studies.

In this research study, the investigators are looking to see if adding NOV-002 to the chemotherapy drug carboplatin works in treating ovarian cancer in women whose cancer has stopped responding to carboplatin chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian, primary peritoneal, or fallopian tube cancer
* ECOG 0-1
* Platinum resistant or refractory disease defined as progressive disease within 6 months of completing or while receiving their last platinum containing regimen
* Measurable disease

Exclusion Criteria:

* History of other malignancies within 2 years except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, incidental stage I endometrial cancer, basal or squamous cell skin cancer
* Major surgery within 2 weeks of study entry
* History of anaphylactic shock with prior platinum chemotherapy
* Known history of central nervous system (CNS) metastases unless subject has had treatment with surgery or radiation therapy and is neurologically stable
* Treatment with more than 3 lines of chemotherapy
* Chronic use of systemic corticosteroids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Kransner, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana Farber Cancer/Partners Cancer Care, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trials opened to enrollment July 2006 and the study was closed out June 2008. Recruitment locations were: Dana Farber Cancer/Partners Cancer Care, Boston, MA and Massachusetts General Hospital, Boston, MA
Pre-assignment Details: Patients were platinum refractory/resistant, with measurable disease and ≤ 3 prior lines.
Period: Overall Study
Arm/Group | NOV-002 Plus Carboplatin
Started | 16 (1 subject enrolled but not treated (off-trial for patient discretion))
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | NOV-002 Plus Carboplatin
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Time Frame: At treatment completion (8 weeks) and monthly until disease progression
Measure: Number; unit: Participants
Arm/Group | NOV-002 Plus Carboplatin
Number analyzed (Participants) | 15
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Stable Disease (SD) | 8
  Progressive Disease (PD) | 6

2. Secondary Outcome: Safety of NOV-002 and Carboplatin
Time Frame: Duration of trial and through 30-day follow-up period after final treatment
Measure: Number; unit: Adverse Events
Arm/Group | NOV-002 Plus Carboplatin
Number analyzed (Participants) | 15
Adverse Events
  CTC Grade 4 Adverse Events | 0
  CTC Grade 3 Adverse Events | 8
  CTC Grade 3 Related Adverse Events | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: From time of treatment start to time of disease progression
Measure: Mean (Full Range); unit: Weeks
Arm/Group | NOV-002 Plus Carboplatin
Number analyzed (Participants) | 15
Weeks | 19.4 [4 to 38]

ADVERSE EVENTS:
Time Frame: Duration of trial (up to 8 weeks) and through 30-day follow-up period after final treatment
Arm/Group | NOV-002 Plus Carboplatin
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NOV-002 Plus Carboplatin (N=15)
Abdominal pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
DVT (Vascular disorders) | 1
Bowel Obstruction (Gastrointestinal disorders) | 1
Platinum Allergy (Immune system disorders) | 2
Depression (Psychiatric disorders) | 1
Syncope (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NOV-002 Plus Carboplatin (N=15)
Lymphopenia (Blood and lymphatic system disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 9
Oedema peripheral (General disorders) | 3
Hypersensitivity (Immune system disorders) | 2
Haemoglobin decreased (Investigations) | 6
Platelet count decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Nervous system disorders (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
The criterion for continuing to Stage II of the study (≥ 2 responses) was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No